CLINICAL TRIAL: NCT05666037
Title: Effectiveness of Interactive Mobile Health Intervention to Improve Early Postpartum Modern Contraceptive Method Uptake Among Women in North East Ethiopia: Community Based Cluster Randomized Control Trial
Brief Title: Interactive Mobile Health Intervention to Improve Early Postpartum Modern Contraceptive Method Uptake
Acronym: EPPMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Niguss Cherie, Assistant professor, Wollo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JUIH/IRB/229/22
Record Dates: First submitted 2022-12-05; First posted 2022-12-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2022-12

CONDITIONS: Other Cardiovascular Diseases of Mother, Postpartum
Keywords: Early post partum, Contraceptive method, Ethiopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive mobile health intervention.
  Interventions: Behavioral: Mobile health intervention(mHealth)
- Control group (No Intervention): The control arm will be received the existed current health delivery approach, not received mobile health sending message service.

INTERVENTIONS:
Behavioral: Mobile health intervention(mHealth) — The intervention group will receive mobile health messaging intervention on behavior change to uptake early postpartum modern contraceptive method.
  Arms: Intervention group

SUMMARY:
The main aim of this study is to determine effectiveness of mobile health intervention to improve early postpartum modern contraceptive service uptake among postpartum women in Dessie and Kombolcha town zones, North east Ethiopia. This study will be conducted in Dessie and Kombolcha zones in Amhara region, North east Ethiopia. The largest sample size will be taken and total sample size will be 784.

DETAILED DESCRIPTION:
The main aim of this study is to determine effectiveness of mobile health intervention to improve early postpartum modern contraceptive service uptake among postpartum women in Dessie and Kombolcha town zones, North east Ethiopia. This study will be conducted in Dessie and Kombolcha zones in Amhara region, North east Ethiopia. The largest sample size will be taken and total sample size will be 784.

Cluster randomized control trial behavioral intervention sampling technique will be deployed. First participants will be grouped in to two arms based on randomization of clusters. The intervention arm will take the new mobile health intervention with existed health care practice and the control arm will take the existed current health care practice. Intervention mobile health messages will be developed from family planning behavior change framework and national guidelines. Data will be collected by using pre-tested interviewer administered structured questionnaires. Data will be collected in four different phases. Open data kit (ODK) will be used for data collection. Duration of intervention will be 4 months. Descriptive analyses will be made by computing proportions and summary statistics. Statistical package to social science (SPSS.26) and STATA.15 soft wares will be used to do analysis. Structural Equation Modeling (SEM) or path analysis will be done to identify the fitted components to determine latent variables.

ELIGIBILITY:
Inclusion Criteria:

All mothers who will be 24-28 week of gestation and have access to mobile phone in the study area will be recruited to this study.

Exclusion Criteria:

* Pregnant women, who will be assumed to have serious medical problems, will be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Early postpartum family planning is outlined as women who have will be used any kind of modern birth control technique at intervals the primary six weeks when she gave birth. | Two weeks after intervention completed the outcome will be measured.
  If the respondent answers yes it will be coded "1" and if not coded as "0"

CONTACTS AND LOCATIONS:
Overall Officials: Niguss Cherie, MPH, Principal Investigator — Wollo Universirty
Locations (1):
- Dessie and Kombolcha, Dessie, South Wollo, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The data will be kept confidential

REFERENCES:
- [Background] Adane M, Cherie N, Damtie Y, Malde M, Chanie MG. Sexual and reproductive health service needs among youths attending preparatory school in Debre Tabor Town, Northwest Ethiopia. SAGE Open Med. 2022 Jul 24;10:20503121221113667. doi: 10.1177/20503121221113667. eCollection 2022. PMID 35910818
- [Derived] Cherie N, Wordofa MA, Debelew GT. Effectiveness of an Interactive Mobile Health Intervention (IMHI) to enhance the adoption of modern contraceptive methods during the early postpartum period among women in Northeast Ethiopia: A cluster Randomized Controlled Trial (RCT). PLoS One. 2024 Nov 14;19(11):e0310124. doi: 10.1371/journal.pone.0310124. eCollection 2024. PMID 39541340